CLINICAL TRIAL: NCT06608303
Title: Study on the Effectiveness and Safety of Topical Human Granulocyte Macrophage Stimulating Factor Gel in the Treatment of Diabetic Wounds During the Granulation Growth Phase
Brief Title: Macrophage Stimulating Factor in the Treatment of Diabetic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2024-Jinfuning
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Wound
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Human Granulocyte Macrophage Stimulating Factor Gel (Experimental): The diabetic wounds were treated with Topical Human Granulocyte Macrophage Stimulating Factor Gel for 2 weeks on top of the standard clinical treatment protocol.
  Interventions: Drug: Topical Human Granulocyte Macrophage Stimulating Factor Gel
- saline (Placebo Comparator): The diabetic wounds were treated with saline for 2 weeks on top of the standard clinical treatment protocol.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Topical Human Granulocyte Macrophage Stimulating Factor Gel — Human granulocyte macrophage colony-stimulating factor (rhGM-CSF), as a multifunctional haematopoietic factor, stimulates the proliferation and differentiation of haematopoietic precursor cells to granulocyte macrophages and promotes their peripheral translocation, as well as enhances phagocytosis and secretion of granulocytes and macrophages [11]. Since macrophages are key players in regulating the inflammatory response of wounds and promoting wound repair, rhGM-CSF is thought to potentially play a positive role in the treatment of acute and chronic wounds.
  Arms: Topical Human Granulocyte Macrophage Stimulating Factor Gel
Drug: Saline (NaCl 0,9 %) (placebo) — placebo
  Arms: saline

SUMMARY:
With the aging of the population, the incidence of diseases such as diabetes, chronic atherosclerotic occlusion, cerebrovascular disease, and cancer is increasing year by year, and has led to an increasing incidence of chronic wounds such as diabetic foot, ischaemic ulcers, venous ulcers, pressure injuries, and radiation ulcers. In addition to the high age and chronic diseases that make the treatment of wounds difficult and long, chronic wounds remain in the proliferative stage, unable to carry out normal repair, which is also an important reason for the prolonged healing of wounds, which seriously affects the quality of life of patients and creates a huge social and family burden. In the United States, chronic hard-to-heal wounds exist in approximately 6.5 million people each year, costing the healthcare system more than $25 billion annually and increasing each year with the increased prevalence of diabetes and other diseases that affect wound healing. How to make chronic wounds heal quickly and well is a huge challenge that affects people's access to health today.

Macrophages are important cells involved in the inflammatory and proliferative phases of wounds, and are thought to play a key role in regulating the inflammatory response of wounds and promoting wound repair and reconstruction. Recombinant human granulocyte macrophage colony-stimulating factor (rhGM-CSF), as a multifunctional haematopoietic factor, can stimulate the proliferation and differentiation of haematopoietic precursor cells to granulocyte macrophage and promote their peripheral transfer, as well as enhance phagocytosis and secretion of granulocytes and macrophages. Therefore rhGM-CSF is thought to have a possible positive role in the treatment of acute and chronic wounds and has been confirmed in several basic and clinical studies.

Topical human granulocyte macrophage stimulating factor gel (JinFuNing), which has been approved and marketed by the state for the treatment of acute and chronic wounds, is able to play a role in promoting wound repair, neovascularisation, and epithelial crawling, and has already achieved a certain degree of efficacy in promoting wound healing. This study accumulates clinical evidence-based medical evidence for more precise use of topical human granulocyte macrophage stimulating factor gel, and explores the clinical efficacy and safety of Jinfuning in the granulation growth phase of diabetic wounds.

DETAILED DESCRIPTION:
2. Approximately 40 people will participate in this study at the Wound Treatment Centre of Peking University Third Hospital.

3. What is included in this study? Study design: prospective, blinded evaluation, randomised controlled study; Inclusion criteria: (1) Subjects aged 18-80 years; (2) Confirmed diagnosis of type 1 or type 2 diabetes mellitus that meets the standard definition of the World Health Organization, with glycaemic control and glycated haemoglobin HbA1c level of less than 10% prior to enrolment; (3) Wound type belonging to the ulcer category; (4) Wound etiology belonging to the diabetic wounds, which are mainly due to the abnormalities of glucose, resulting in poor or prolonged healing, and needing to undergo standard wound treatment; (5) the wound staging was in the granulation growth phase; (6) voluntary participation in this study and signing the informed consent.

Exclusion criteria: (1) severe diseases such as acute infarction, heart failure, hepatitis, shock, and expiratory failure, which had not been corrected; (2) uncontrolled blood glucose, fasting blood glucose > 15 mmol/L and glycated haemoglobin > 12%; (3) active bleeding within the wound, which could not be carried out with the conventional basic treatment regimen; (4) serum albumin < 20 g/L; haemoglobin < 60 g/L; platelets < 50×109 /L; (5) disseminated infection status, being treated or about to be treated with antibiotics; (6) subjects with advanced malignancy; (7) active autoimmune disease; (8) previous allergy to bioactive glass ointment dressings (autogenous); (9) subjects who are unable to cooperate or mentally challenged; (10) subjects who, in the judgement of the investigator, have a clearly unremovable cause of affecting wound healing that is unsuitable for this study or unable to comply with the requirements of this study.

Randomisation to groups was based on the staging of chronic wounds and only after the stage conditions were met.

of granulation, divided into: 20 cases in the control group and 20 cases in the treatment group.

You will be randomly assigned (like a coin flip) to either group, with a 50% chance of being assigned to the control group; the chance of being assigned to the treatment group is a 50% chance of being assigned to the treatment group. Treatment Except for the use of topical human granulocyte macrophage stimulating factor gel, the treatment and examination protocols will be consistent with the standard clinical protocols for the control group, including, but not limited to, strict glycemic control, antihypertensive, lipid-lowering, improvement of microcirculation, anti-infective, nutritive neurological, systemic nutritional support, local physiotherapy, arterial intraluminal shaping, debridement, dead bone removal, tendon probing and resection, and negative pressure therapy.

The study steps are as follows:

1. Perform wound photography, wound area measurement and recording, and complete wound bed preparation (wound hygiene, effective debridement);
2. Apply topical human granulocyte macrophage stimulating factor gel treatment:

   Control group: clinical standard treatment protocol; Treatment group: on the basis of the clinical standard treatment protocol, use topical human granulocyte macrophage stimulating factor gel to treat the wound for 2 weeks, applied to the wound with a thickness of 2 mm. if possible, on the 7th-14th day after the application of the drug, the debridement waste tissue will be sent for examination, and improve the transcriptome (Bulk RNA-seq) analysis and detection, or other proteins, gene detection and immunofluorescence, etc. after the examination in accordance with the medical treatment. Dispose of the tissue as medical waste.
3. Clinical standard treatment plan For each wound, according to the wound status, stage, size, etiology and location, the optimal treatment plan and necessary surgical treatment measures are selected in accordance with clinical diagnosis and treatment routines, including but not limited to strict control of blood glucose, lowering blood pressure, lowering lipids, improvement of microcirculation, anti-infections, nutritional neurotoxicity, systemic nutritional support, local physiotherapy, arterial endoluminal shaping, debridement, dead bone removal, tendon probing and resection, and negative pressure treatment.

Note: Although the general principles of wound treatment are usually the same, due to the variety of wound status, stage, size, etiology, and location, each treatment plan must be tailored to address individualised problems in order to achieve a more effective wound repair, and even then, with the current technological capabilities of mankind, some wounds will still have delayed healing or non-healing. Therefore, clinical observations must be based on standard treatment protocols in order to minimise additional factors affecting wound repair.

This is a prospective, blinded evaluation, randomised controlled study and you may be randomly assigned to either the control or observation group. You will know exactly which group you are in, whether or not you are applying topical human granulocyte macrophage stimulating factor gel, and you will be able to observe the healing process of your wound together.

4. How long will this study last? You participate in this study for 3 weeks, with follow-up records to be completed on the day of treatment (Day 0), Week 1 after treatment (Day 7), Week 2 after treatment (Day 14), and Week 3 after treatment (Day 21). Wound area changes and safety indicators are observed at weekly follow-up visits. Your regular follow-up appointments and medication changes will be our follow-up visits, and will not add to the number of additional visits or costs if there are no special circumstances.

You may choose to leave the study at any time without losing any of the benefits you would otherwise receive. However, if you decide to leave the study during the course of the study, a check-up may be carried out after the withdrawal, if necessary, to take into account your safety concerns.

5. What are the risks of participating in this study? All subjects eligible for enrolment have chronic ulcer type wounds. The wounds must all be rigorously prepared and the protocol will only be administered after your general condition has improved. At this point, you are enrolled in treatment and your overall risk is already low.

In this study, the investigators have added topical human granulocyte macrophage-stimulating factor gel to the optimal clinical regimen for the wounds in the Jinfuning group, but the rest of the treatment is routine. The optimal clinical regimen has been in place for several years and has been stable and reliable, and has cured a large number of people. However, by joining this study, it does not mean that you are guaranteed to be treated with Topical Human Granulocyte Macrophage Stimulating Factor (HMMSF) Gel, and there is a 50% chance you will be given the Topical HMMSF Gel regimen.

Topical human granulocyte macrophage stimulating factor gel mainly promotes the proliferation and differentiation of granulocyte macrophages, improves the inflammatory state, secretes a variety of wound repair proteins and factors, and promotes the proliferation and repair of wounds, non-local antimicrobial agents, and the main risk of topical application is the occurrence of disseminated infection. Strict wound hygiene, effective bacterial reduction and debridement, and the use of local antimicrobial agents must be carried out before application to minimise the risk of infection. The patients enrolled in this trial were all patients with systemic infection or disseminated infection that had been controlled and entered the period of granulation growth, and the local application of topical human granulocyte macrophage stimulating factor gel was conducive to accelerating the formation of new microvessels and the growth of local granulation tissues, and the frequency of dressing changes was sufficient, so that timely intervention could be made once signs of disseminated infection were detected, and the clinic routinely had a series of measures to control the dissemination of infections.

Secondly, allergic reaction to topical human granulocyte macrophage stimulating factor gel. After applying the dressing, each patient was observed for 10-30 minutes without discomfort before being allowed to leave the hospital, and the patient was told to return to the hospital if he/she felt unwell. Each time the dressing is opened, the wound oozing and the surrounding skin should be observed for allergic reactions such as rash and redness. If an allergic reaction occurs, different anti-allergic treatments will be given depending on the severity.

Of course, diabetic wounds are a worldwide problem with diverse etiologies, and even with topical human granulocyte macrophage stimulating factor gel treatment, they may still not heal. In addition, participants' co-morbidities will not get better with Topical Human Granulocyte Macrophage Stimulating Factor Gel treatment. If participants have multi-system diseases, please take the medication on time to ensure that participants' condition is stable, and if there is a progression of participants' co-morbidities, please go to the appropriate department in time for treatment.

If participants have an adverse reaction, the study doctor will terminate the study depending on the severity.

6. What are the benefits of participating in the study? If the participants agree to participate in this study, it is possible that the participants may have a benefit from wound treatment, but the investigators cannot guarantee that participants will have such a benefit. The investigators hope that the information gained from participants' participation in this study will benefit the participants and other patients with the same condition in the future.

7. What other medical options are available? If the participants do not take part in this study, participants will have conventional wound treatment. If participants participate in this study, there is a 50% chance that participants will be treated with topical human granulocyte macrophage stimulating factor gel in addition to participants' regular treatment.

8. Will my information be kept confidential? The investigators will keep participants' study records confidential as required by law. Our laws provide for privacy, data and security of authorised access. Participants' information will be de-identified in this study, the investigators will represent participants with a unique number, and their information will not be transferred to a third party. Waste tissue specimens collected for this study will also be de-identified and destroyed after testing. Their identity will not be disclosed when the research information and data obtained from this study are presented at scientific meetings or in scientific journals. However, their records may be reviewed to ensure that the study complies with applicable laws and regulations. The reviewers will include the relevant national regulatory authorities and the Ethics Committee of the Third Hospital of Peking University. Participants have the right to withdraw from this study at any time. If participants withdraw, the information already collected will not be used for this study, and after withdrawal, no more information related to the study will be collected.

9. What about the cost of the study? The treatment group needs to be treated with topical human granulocyte macrophage stimulating factor gel, which will be provided by the drug manufacturer free of charge during the trial period. Wound assessment, information collection, wound dressing changes, examination and test items, and follow-up visits are routine clinical practice.

10. What compensation will I receive? This study does not increase the cost of routine care and is not compensated.

11. If a study-related injury occurs If participants suffer an injury as a result of their participation in the study, Peking University Third Hospital will provide the necessary medical care and, in accordance with applicable laws and regulations, will cover the costs of direct treatment and appropriate compensation.

12. Refusing to participate or withdrawing from the study Participation in the trial is voluntary and participants may refuse to participate or withdraw from the trial in any way at any stage of the trial without discrimination or retaliation, and your medical treatment and rights will not be affected.

If participants have a serious adverse reaction, or if their study doctor feels that it is not in their best interest to continue in the study, he/she may decide to withdraw participants from the study. Participants will be notified promptly if this happens and their study doctor will discuss the other options participants have with you. If their doctor feels that an abrupt discontinuation of the trial will affect your health, he/she may ask participants to come to the hospital for a check-up before stopping the trial.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of type 1 or type 2 diabetes mellitus that meets the standard World Health Organization definition, with blood glucose controlled prior to enrolment and a glycated haemoglobin HbA1c level of less than 10%;
* the type of wound is an ulcer;
* the wound etiology is diabetic, mainly abnormalities in blood glucose, resulting in poor or prolonged healing and requiring standard wound therapy;
* the staging of the wound is in the granulation phase;
* voluntary participation in the study and signing of an informed consent form.

Exclusion Criteria:

* acute heart attack, heart failure, hepatitis, shock, expiratory failure and other serious diseases that have not been corrected;
* uncontrolled blood glucose, fasting blood glucose > 15 mmol/L and glycated haemoglobin > 12%;
* active bleeding in the wound, which does not allow the implementation of the conventional basic treatment plan;
* serum albumin < 20 g/L; haemoglobin < 60 g/L; platelets < 50 x 109/L;
* a state of disseminated infection that is being or will be treated with antibiotics
* patients with advanced malignant tumours;
* active autoimmune disease;
* previous allergy to topical human granulocyte macrophage stimulating factor gel (Jinfuning);
* inability of the patient to co-operate or mental disorder;
* in the judgement of the investigator, the subject has a clearly irremovable cause of wound healing, is unsuitable for the study or is unable to comply with the requirements of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
wound area reduction rate | From enrollment to the end of treatment at 2 weeks
  Pre-treatment area minus post-treatment area, then divided by pre-treatment area

SECONDARY OUTCOMES:
wound healing rate | From enrollment to the end of treatment at 2 weeks
  Percentage of healed wounds to total cases by D14
Granulation tissue status | From enrollment to the end of treatment at 2 weeks
  They were classified as healthy granulation, inflammatory granulation, infected granulation, oedematous granulation, and aged granulation. D0/D14, wound granulation tissue status was recorded separately
wound infection control | From enrollment to the end of treatment at 2 weeks
  0 points for no infection, 1 point for reduction of localised infection; 2 points for maintenance or exacerbation of localised infection; 3 points for disseminated infection; record D0/D14, the status of the wound infection and record the scoring results respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No